CLINICAL TRIAL: NCT00770913
Title: Double-blind Comparative Study of E3810 Tablets (10 or 20 mg b.i.d.) to Evaluate Efficacy and Safety in Patients With Refractory Reflux Esophagitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E3810-J081-304
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2012-04-13 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2010-06

CONDITIONS: Refractory Reflux Esophagitis
Keywords: reflux esophagitis; rabeprazole; GERD; Japan
MeSH Terms: conditions — Esophagitis, Peptic; Gastroesophageal Reflux | interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: E3810
- 2 (Experimental)
  Interventions: Drug: E3810
- 3 (Experimental)
  Interventions: Drug: E3810

INTERVENTIONS:
Drug: E3810 — 20 mg taken orally, once a day for 8 weeks.
  Other Names: Aciphex
  Arms: 1
Drug: E3810 — 10 mg, taken orally, twice a day for 8 weeks.
  Other Names: Aciphex
  Arms: 2
Drug: E3810 — 20 mg taken orally, twice a day for 8 weeks.
  Other Names: Aciphex
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of E3810 tablets in patients with Proton Pump Inhibitor-resistant reflux esophagitis.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blinded study. The efficacy with E3810 20 mg once daily is compared with E3810 20 mg twice daily and 10 mg twice daily using endoscopic recovery. The frequency of adverse event, etc., will be compared among 3 groups for safety assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have mucosal breaks (erosions, ulcers) on endoscopy and are diagnosed with reflux esophagitis.
* Proton Pump Inhibitor standard dose-resistant reflux esophagitis.
* Patients who are 20 years and older when informed consent is obtained.

Exclusion Criteria:

* Patients with a concurrent severe illness, serious heart disease, comorbid severe disease such as hematology, kidney disease, or liver disease.
* Patients with malignancy.
* Patients who are taking another trial drug or the interval between the end of treatment and screening is less than 12 weeks.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2008-10; Primary Completion 2009-11 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomoki Kubota, Study Director — New Product Development Dept., Clinical Research Center
Locations (54):
- Japan (54):
  - Nagakute, Aichi-ken
  - Nagoya, Aichi-ken
  - Akita, Akita
  - Abiko, Chiba
  - Kashiwa, Chiba
  - Yachiyo, Chiba
  - Chikushino-shi, Fukuoka
  - Fukuoka, Fukuoka
  - Omuta, Fukuoka
  - Tagawa, Fukuoka
  - Kōriyama, Fukushima
  - Gifu, Gifu
  - Hashima, Gifu
  - Maebashi, Gunma
  - Hiroshima, Hiroshima
  - Asahikawa, Hokkaido
  - Sapporo, Hokkaido
  - Itami, Hyōgo
  - Nishinomiya, Hyōgo
  - Hitachi, Ibaraki
  - Takamatsu, Kagawa-ken
  - Kagoshima, Kagoshima-ken
  - Kirishima, Kagoshima-ken
  - Kawasaki, Kanagawa
  - Yokohama, Kanagawa
  - Kochi, Kochi
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Ishinomaki, Miyagi
  - Nagasaki, Nagasaki
  - Yamatokōriyama, Nara
  - Beppu, Oita Prefecture
  - Ōita, Oita Prefecture
  - Okayama, Okayama-ken
  - Hirakata, Osaka
  - Osaka, Osaka
  - Karatsu, Saga-ken
  - Saga, Saga-ken
  - Kusatsu, Shiga
  - Izumo, Shimane
  - Matsue, Shimane
  - Fujieda, Shizuoka
  - Hamamatsu, Shizuoka
  - Shimada, Shizuoka
  - Shizuoka, Shizuoka
  - Ohtawara, Tochigi
  - Bunkyo, Tokyo
  - Setagaya City, Tokyo
  - Shinagawa, Tokyo
  - Shinjuku, Tokyo
  - tabashi City, Tokyo
  - Yamagata, Yamagata
  - Hōfu, Yamaguchi
  - Shimonoseki, Yamaguchi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 71 centers in Japan during the period of 17-Oct-2008 to 12-Nov-2009.
Pre-assignment Details: There was no run-in phase before assignment to E3810 treatment groups in this study.
Groups:
- E3810 20 mg Once Daily: E3810 20mg once daily orally for 8 weeks
- E3810 10 mg Twice Daily: E3810 10mg twice daily orally for 8 weeks
- E3810 20 mg Twice Daily: E3810 20mg twice daily orally for 8 weeks
Period: Overall Study
Arm/Group | E3810 20 mg Once Daily | E3810 10 mg Twice Daily | E3810 20 mg Twice Daily
Started | 113 | 111 | 113
Completed | 102 | 103 | 100
Not Completed | 11 | 8 | 13
Not completed — Adverse Event | 1 | 3 | 6
Not completed — Refusal to continue participation | 6 | 4 | 5
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Protocol Violation | 3 | 0 | 1
Not completed — Incorrect drug was allocated | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E3810 20 mg Once Daily | E3810 10 mg Twice Daily | E3810 20 mg Twice Daily | Total
Number analyzed (Participants) | 110 | 111 | 111 | 332
Age Continuous [Mean (Standard Deviation); unit: years] — Full Analysis Population
  years | 64.5 (13.9) | 65.5 (13.3) | 66.6 (13.8) | 65.5 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 59 | 62 | 174
  Male | 57 | 52 | 49 | 158
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 110 | 111 | 111 | 332

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Healing Demonstrated Via Upper Gastrointestinal Endoscopy (Modified Los Angeles Classification: Grade N)
Description: Grade N indicates a normal appearance of lower esophageal mucosa
Time Frame: 8 weeks
Population: The primary analysis was on the full analysis set (FAS) population.
Measure: Number; unit: Percentage of Participants
Groups:
- E3810 20 mg Once Daily: E3810 20 mg once daily orally for 8 weeks
- E3810 10 mg Twice Daily: E3810 10 mg twice daily orally for 8 weeks
- E3810 20 mg: E3810 20 mg twice daily orally for 8 weeks
Arm/Group | E3810 20 mg Once Daily | E3810 10 mg Twice Daily | E3810 20 mg
Number analyzed (Participants) | 113 | 111 | 113
Percentage of Participants | 58.8 | 78.4 | 77.0

ADVERSE EVENTS:
Description: The safety population includes all participants who took at least one dose of the assigned intervention. No.of Participants Analyzed: 113, 111, 113.Participants affected/at risk: 112, 111, 114. The drug was incorrectly prescribed. It should have been 20mg twice daily, but 20mg once daily was mistakenly prescribed despite of correct allocation.
Arm/Group | E3810 20 mg Once Daily | E3810 10 mg Twice Daily | E3810 20 mg
Serious Adverse Events (participants affected / at risk) | 3/112 | 6/111 | 5/114
Other Adverse Events (participants affected / at risk) | 27/112 | 25/111 | 20/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E3810 20 mg Once Daily (N=112) | E3810 10 mg Twice Daily (N=111) | E3810 20 mg (N=114)
Cellulitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 1 | 0 | 0
Putamen haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E3810 20 mg Once Daily (N=112) | E3810 10 mg Twice Daily (N=111) | E3810 20 mg (N=114)
Nasopharyngitis (Infections and infestations) | 8 | 7 | 4
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2
Constipation (Gastrointestinal disorders) | 2 | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 3 | 7 | 7
Blood triglycerides increased (Investigations) | 5 | 1 | 1

LIMITATIONS AND CAVEATS:
In the Participant flow section, there is only one "Reason for Not Completed" per participant reported, even if there were multiple reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No